CLINICAL TRIAL: NCT07280000
Title: The Effect of the Action Plan Developed Within the Framework of Respectful Maternity Care in Postpartum Care on Maternal and Neonatal Outcomes
Brief Title: Effect of a Respectful Maternity Care-Based Action Plan in Postpartum Care on Maternal and Neonatal Outcomes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ilayda sel (Other)
Responsible Party: Sponsor-Investigator, ilayda sel, Research Assistant (Women Health and Diseases Nursing), Bandırma Onyedi Eylül University
Organization: Bandırma Onyedi Eylül University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ISB-WH-02
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Postpartum Care; Maternal Health Care; Newborn Health; Postpartum Depression (PPD); Breastfeeding; Quality of Care; Maternal Satisfaction
Keywords: Respectful Maternity Care; Postpartum Care; Maternal Health; Newborn Health
MeSH Terms: conditions — Depression, Postpartum; Breast Feeding

STUDY DESIGN:
Intervention Model Description: This is a quasi-experimental, controlled before-after study with two parallel groups. Postpartum women receiving routine care before the training and action plan implementation constitute the control group, and postpartum women receiving care after the intervention constitute the intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control: Routine Postpartum Care (No Intervention): Participants in this arm will receive routine postpartum care practices currently provided at the study site, without exposure to the respectful maternity care training or action plan components. Usual clinical care protocols and standard postpartum follow-up procedures will be applied.
- Intervention: Respectful Maternity Care Action Plan (Experimental): Participants in this arm will receive postpartum care delivered by nurses and midwives trained in the Respectful Maternity Care (RMC) Action Plan. The intervention includes structured training for postpartum professionals, implementation of evidence-based respectful maternity practices, and application of the developed RMC program content and postpartum care forms. Care will emphasize dignity, privacy, informed consent, emotional support, newborn bonding, breastfeeding support, and person-centered communication.
  Interventions: Behavioral: Respectful Maternity Care Training and Action Plan

INTERVENTIONS:
Behavioral: Respectful Maternity Care Training and Action Plan — This intervention involves a structured Respectful Maternity Care (RMC) training program for nurses and midwives, followed by the implementation of an evidence-based RMC action plan during postpartum care. The training includes modules on dignity, privacy, informed consent, effective communication, emotional support, newborn bonding and breastfeeding support, and person-centered postpartum practices. Participants in the intervention arm will receive postpartum care according to the RMC guidelines and structured care forms developed for the study.
  Arms: Intervention: Respectful Maternity Care Action Plan

SUMMARY:
This study will examine whether a Respectful Maternity Care-based action plan can improve the quality of postpartum care and maternal and newborn outcomes. Nurses and midwives will receive a three-day interactive training about respectful, evidence-based postpartum care. After training, a unit-level action plan will be implemented, including supportive visits, educational materials, and feedback meetings. Women receiving routine postpartum care before the intervention will be compared with women receiving care after implementation. Outcomes will include respectful maternity care experiences, maternal satisfaction, exclusive breastfeeding at 6-8 weeks, maternal mental health, mother-infant bonding, and postpartum complications. The goal of this study is to promote respectful, high-quality postpartum care and improve the health and well-being of mothers and newborns.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women aged 18 years and older
* Gave birth at 37-42 gestational weeks (vaginal or cesarean)
* Have a single, healthy newborn
* No chronic medical conditions
* No history of high-risk pregnancy or fetal complications
* No communication barriers (e.g., visual or hearing impairment)
* Able to speak and understand Turkish
* Literate and able to read and write in Turkish

Exclusion Criteria:

* Development of maternal or neonatal complications during the postpartum follow-up period
* Inability to reach the mother at the 8-week postpartum follow-up

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study includes postpartum individuals who are biologically female.
Enrollment: 500 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Respectful Maternity Care Score | Baseline (within 24 hours postpartum) and 6 weeks postpartum
  Respectful maternity care will be assessed using the Respectful Maternity Care (RMC) scale, which evaluates dignity, privacy, informed consent, emotional support, communication, and person-centered postpartum practices. Higher scores indicate higher levels of respectful maternity care.

SECONDARY OUTCOMES:
Maternal Satisfaction with Postpartum Care | At discharge (within 48 hours postpartum)
  Maternal satisfaction with postpartum care will be assessed using a validated postpartum satisfaction questionnaire, measuring perceptions of communication, emotional support, involvement in care, and overall satisfaction with hospital postpartum services. Higher scores indicate greater satisfaction.
Postpartum Depression Score | 6 weeks postpartum
  Depressive symptoms will be evaluated using the Edinburgh Postpartum Depression Scale (EPDS). Higher scores indicate higher depressive symptoms. A cutoff score of ≥13 suggests risk of postpartum depression.
Adherence to Evidence-Based Postpartum Care Practices | Immediately postpartum (within 24 hours)
  A structured postpartum care checklist will be used to evaluate compliance with respectful and evidence-based postpartum care practices (privacy, informed consent, emotional support, newborn bonding, breastfeeding support, early mobilization, postpartum monitoring). Higher scores indicate greater adherence to evidence-based guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: İlayda Sel Bilim, MSc, RN, Principal Investigator — Istanbul University - Cerrahpasa; İlkay Güngör Satılmış, Prof., Study Chair — Istanbul University - Cerrahpasa
Locations (1):
- Bakırköy Dr. Sadi Konuk Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No, individual participant data (IPD) will not be shared. Due to ethical considerations and the sensitive nature of maternal and postpartum health data, participant confidentiality will be strictly protected. Only aggregated results will be published, and data access will remain restricted to the study team in accordance with ethical approval.

REFERENCES:
- [Result] Bohren MA, Vogel JP, Hunter EC, Lutsiv O, Makh SK, Souza JP, Aguiar C, Saraiva Coneglian F, Diniz AL, Tuncalp O, Javadi D, Oladapo OT, Khosla R, Hindin MJ, Gulmezoglu AM. The Mistreatment of Women during Childbirth in Health Facilities Globally: A Mixed-Methods Systematic Review. PLoS Med. 2015 Jun 30;12(6):e1001847; discussion e1001847. doi: 10.1371/journal.pmed.1001847. eCollection 2015 Jun. PMID 26126110